CLINICAL TRIAL: NCT05663736
Title: Comparison in Effect of Gemigliptin Versus Glimepiride on Cardiac Diastolic Function in Patients With Type 2 Diabetes Uncontrolled With Metformin
Brief Title: Effect of Gemigliptin Versus Glimepiride on Cardiac Diastolic Function in Patients With Type 2 Diabetes
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Soo Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B-1712/438-004
Record Dates: First submitted 2022-12-15; First posted 2022-12-23 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Ejection Fraction
MeSH Terms: interventions — LC15-0444; glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gemiglipitin (Experimental): A DPP4 inhibitor gemigliptin treatment group
  Interventions: Drug: Gemigliptin
- Glimepiride (Active Comparator): A sulfonylurea glimepiride treatment group
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: Gemigliptin — DPP-4 inhibitor
  Other Names: Zemiglo
  Arms: Gemiglipitin
Drug: Glimepiride — Glimepiride
  Arms: Glimepiride

SUMMARY:
Among DPP-4 inhibitors, gemigliptin is a relatively recently developed drug, and many clinical studies have shown results that are equivalent to or superior to existing DPP-4 inhibitors such as sitagliptin. However, studies on the safety of gemigliptin in cardiovascular disease have not been conducted, and studies on its effect on cardiac function are lacking. Considering the increase in hospitalizations due to heart failure found in some DPP-4 inhibitor studies, investigation of directly effect of gemigliptin on heart function would be clinically important.

DETAILED DESCRIPTION:
Many international guidelines including the American Diabetes Association and Korean diabetes association recommend metformin as an initial hypoglycemic agent. They also suggest early active treatment for patients with type 2 diabetes (T2D) when it is difficult to reach the target blood sugar with metformin monotherapy alone. This is a strategy to minimize the period of exposure to hyperglycemia. However, when choosing the second agent, both efficacy and safety should be considered.

The American Diabetes Association guidelines recommend to using glucagon-like peptide 1 receptor agonist (GLP-1 RAs) for patients with T2D at high atherosclerotic cardiovascular disease and sodium-glucose cotransporter-2 inhibitor for T2D patients at high risk of heart failure or chronic kidney disease. However, people at this condition are not majority in many countries.

Sulfonylurea is an oral hypoglycemic agent that was first developed in the 1950s and has been widely used for a long time. Since these sulfonylureas are complementary to metformin in their mechanism of action, sulfonylureas and metformin are one of the suitable combination therapies. In fact, in a phase 3 clinical study conducted on Koreans, compared to increasing the dose of metformin, combined administration of glimepiride and metformin proved superior in the hypoglycemic effect. However, when glimepiride and metformin were combined, hypoglycemia occurred more frequently than metformin monotherapy, and there was a side effect of weight gain. Therefore, although sulfonylurea and metformin combination therapy is an effective combination in terms of lowering blood sugar, there are doubts as to whether it is the optimal combination therapy due to side effects such as hypoglycemia and weight gain, which are disadvantages of sulfonylurea itself.

Dipeptidyl peptidase-4 (DPP-4) inhibitors are an incretin-based therapy that have proven their hypoglycemic effect in both monotherapy and metformin combination therapy. According to the incretin-based mechanism of action, the risk of hypoglycemia is low, and the weight is neutral with DPP-4 inhibitors. In addition, it can be used without serious adverse events. On the contrary to most GLP-1 RAs, DPP-4 inhibitors are oral antidiabetic agents, which are convenient for physicians to prescribe as well as for patients to take. Of note, this class has been known to be more beneficial in Asian ethnic groups. Thus, DPP-4 inhibitors have been widely used in this region.

Like sulfonylurea, when used in combination with initial metformin, it has a superior blood sugar lowering effect compared to metformin alone. However, when metformin is combined with a DPP-4 inhibitor, the risk of hypoglycemia does not increase unlike when sulfonylurea is combined. Therefore, considering the safety related to the occurrence of hypoglycemia, the DPP-4 inhibitor and metformin combination therapy may be the preferred choice over the sulfonylurea and metformin combination therapy. In several phase 3 studies and registry studies in patients with T2D who failed metformin monotherapy, the addition of a DPP-4 inhibitor to metformin was proven to be safe in hypoglycemia compared to the addition of a sulfonylurea.

Among DPP-4 inhibitors, gemigliptin is a relatively recently developed drug, and many clinical studies have shown results that are equivalent to or superior to existing DPP-4 inhibitors such as sitagliptin. However, studies on the safety of gemigliptin in cardiovascular disease have not been conducted, and studies on its effect on cardiac function are lacking. Considering the increase in hospitalizations due to heart failure found in some DPP-4 inhibitor studies, investigation of directly effect of gemigliptin on heart function would be clinically important.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with type 2 diabetes were eligible if they were aged >20 years, had received metformin (500 mg - 2550 mg) alone for more than 6 weeks and have a glycated hemoglobin of 7%-9.5%.

Exclusion Criteria:

* if they had type 1 diabetes, were pregnant or lactating, or had New York Heart Association class III or IV heart failure. Other exclusion criteria were thyroid stimulating hormone > 10.0 IU/ml, severe infection, chronic kidney disease with eGFR < 30, AST/ALT exceeding 3 times the upper limit of the normal range, use of anti-obesity drugs within 12 weeks of the study, primary coronary intervention for acute coronary syndrome or myocardial infarction within 6 months prior to the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 24 weeks
  Glycated hemoglobin

SECONDARY OUTCOMES:
Ejection fraction | 24 weeks
  Cardiac function
E/e' | 24 weeks
  Cardiac systolic function
LV mass index | 24 weeks
  Cardiac function
LV end-diastolic volumn | 24 weeks
  Cardiac function
NT-proBNP | 24 weeks
  Cardiac biomarker
hsCRP | 24 weeks
  Cardiac biomarker
Adiponectin | 24 weeks
  Metabolic biomarker
Resistin | 24 weeks
  Metabolic biomarker
Troponin I | 24 weeks
  Metabolic biomarker
CK-MB | 24 weeks
  Metabolic biomarker

CONTACTS AND LOCATIONS:
Overall Officials: Soo Lim, MD, Principal Investigator — SNUBH
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No